CLINICAL TRIAL: NCT01089348
Title: Phase II Multicentered Randomized Open-label Study of Effectiveness and Safety of Lactofiltrum in Women With Bacterial Vaginosis
Brief Title: A Pilot Open-label Randomized Study of Lactofiltrum in Women With Bacterial Vaginosis
Acronym: LF-BV-09
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Avva Rus, JSC (Industry)
Collaborators: Kirov State Medical Academy (Unknown); Kirov Regional clinical Center of Perinatology (Unknown)
Responsible Party: Prof. Sergey Dvoryanskiy, Kirov State Medical Academy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 02/09-AVVA RUS
Record Dates: First submitted 2010-03-17; First posted 2010-03-18 (Estimated); Last update posted 2010-07-21 (Estimated); Status verified 2010-07

CONDITIONS: Bacterial Vaginosis
Keywords: Vaginosis, Bacterial; Prebiotics; Lactofiltrum; Therapy
MeSH Terms: conditions — Vaginosis, Bacterial | interventions — Metronidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lactofiltrum (Experimental)
  Interventions: Drug: Lactofiltrum + Metronidazole
- Control (Active Comparator)
  Interventions: Drug: Metronidazole

INTERVENTIONS:
Drug: Lactofiltrum + Metronidazole — Metronidazole 500 mg 1 tablet BID for 7 days + Lactofiltrum 2 tablets 3 times per day for 14 days per os
  Arms: Lactofiltrum
Drug: Metronidazole — Metronidazole 500 mg 1 tablet BID for 7 days per os
  Arms: Control

SUMMARY:
This is a phase II multicenter randomized open-label clinical study that will determine whether treatment with Lactofiltrum (orally administered tablets) in combination with antibiotic therapy (metronidazole) is effective in women with bacterial vaginosis. Lactofiltrum is a composite drug that includes enterosorbent lignin and prebiotic Lactulose. It's supposed that supplement of Lactofiltrum to a standard therapy of bacterial vaginosis (metronidazole administered orally) improves women's general state, leads to better recovery of clinical, microbiological, biochemical and histological features of the disease.

ELIGIBILITY:
Inclusion Criteria:

* bacterial vaginosis.

Exclusion Criteria:

* pregnancy and breast-feeding;
* concomitant infection diseases;
* systemic or topical treatment with antibiotics, steroids, immunosuppressive, cytostatic or antimetabolite agents by the time of inclusion;
* application of intravaginal medicines during participation in the study;
* severe diseases;
* renal and hepatic failure;
* application of pre-, probiotics and antibiotics 2 weeks before inclusion or during participation in the study;
* participation in other clinical study 1 month before inclusion or during participation in the proposed study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2010-07; Primary Completion 2010-10 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Self-reported complaints | Days 0, 14 and 44 after start of intervention
  It's measured by seven ordinal (analog) scales (vaginal itch, vaginal burning, itch of external genitals, burning of external genitals, vaginal discharge, urination disorder,painful intercourse) with minimal value "0" (absent of the complaint-related discomfort) and maximal value "10" (maximal discomfort).

SECONDARY OUTCOMES:
Gynaecological examination | Days 0, 14 and 44 after start of intervention
  It's represented by three ordinal scales with minimal value "0" ("not at all") and maximal value "3" ("severe"). They are measured by physician.
Microscopy of vaginal discharge | Days 0, 14 and 44 after start of intervention
Microbiological examination of vaginal discharge | Days 0, 14 and 44 after start of intervention
pH-test of vaginal discharge | Days 0, 14 and 44 after start of intervention
Microbiological feces analysis | Days 0, 14 and 44 after start of intervention
Blood test | Days 0, 14 and 44 after start of intervention
Urine test | Days 0, 14 and 44 after start of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Lyudmila Kobeleva, MD, PhD, Study Director — Avva Rus, JSC; Sergey Dvoryanskiy, MD, DrSc, Principal Investigator — Kirov State Medical Academy
Locations (2):
- Russia (2):
  - Kirov State Medical Academy, Kirov, Kirov Oblast
  - Kirov Regional Clinical Center of Perinatology, Kirov, Kirov Oblast